CLINICAL TRIAL: NCT04171713
Title: Compared Effects of Mindfulness and Compassion-based Programs on Food Behavior of Patients With Weight Regulation After Bariatric Surgery: a Controlled and Randomized Study
Brief Title: Mindfulness and Compassion-based Programs on Food Behavior of Patients With Weight Regain After Bariatric Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Mente Aberta de Mindfulness (Other)
Responsible Party: Principal Investigator, Marcelo Demarzo, MD, PhD, MD, PhD, Centro Mente Aberta de Mindfulness
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Mindfulness e reganho de peso
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Obesity
Keywords: bariatric surgery; weight regain; food behavior; mindfulness; compassion; empathy
MeSH Terms: conditions — Obesity | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Grup 1 (Experimental): MBHP protocol + TAU
  Interventions: Behavioral: Mindfulness-Based Health Promotion + Treatment as usual; Behavioral: Treatment as usual
- Grup 2 (Experimental): ABCT protocol + TAU
  Interventions: Behavioral: Attachment-based compassion therapy + Treatment as usual; Behavioral: Treatment as usual
- Grup 3 (Active Comparator): TAU
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Mindfulness-Based Health Promotion + Treatment as usual — Structured and developed over eight weeks (8 sessions), participants meet weekly for an average of 2 hours to experience the techniques and conceptual learning about mindfulness and can be adapted to one or 1.5 hour sessions. to be applicable within the contexts of health, education, and organizations. Plus participation in support groups offered by the bariatric surgery clinic with capacity for 40 participants, monthly attendance and duration of 2 hours. In these meetings, there is always the presence of a surgeon, a psychologist and another invited professional (endocrinologist, nutritionist, speech therapist or dentist), who give a thematic lecture and then there is the opening space for doubts and exchange of experiences.
  Other Names: MBHP + TAU
  Arms: Grup 1
Behavioral: Attachment-based compassion therapy + Treatment as usual — It is a program based on one of the fundamental psychological constructs that explain individuals' interpersonal relationships, attachment styles. It lasts 8 weeks in which participants meet for 2 or 2.5 hours at each meeting.
  Other Names: ABCT + TAU
  Arms: Grup 2
Behavioral: Treatment as usual — participation in support groups offered by the bariatric surgery clinic with capacity for 40 participants, monthly attendance and duration of 2 hours. In these meetings, there is always the presence of a surgeon, a psychologist and another invited professional (endocrinologist, nutritionist, speech therapist or dentist), who give a thematic lecture and then there is the opening space for doubts and exchange of experiences.
  Other Names: TAU

SUMMARY:
Weight regain in patients after bariatric surgery has been reported as one of the main failure factors of these surgeries, has important health consequences, such as the return of associated comorbidities, and, until that moment, needs effective treatment. Among its probable causes is the maintenance of dysfunctional eating behavior, even after the procedure. In this context, contemporary, evidence-based mindfulness training protocols focusing on health promotion and socio-emotional skills (compassionate training) have the potential to assist in self-regulation of eating behavior, reducing eating. dysfunctional and facilitating weight self-management. The aim of this study is to compare the preliminary efficacy and feasibility of the Mindfulness-Based Health Promotion (MBHP) and Attachment-Based Compassion Therapy (ABCT) programs in the eating behavior of post-weight regained bariatric patients. The study will be divided into two phases: a cross-analytical study with patients who underwent bariatric surgery between 2012 and 2016, and a controlled and randomized study only with those who obtained weight regain, with mixed data collection. Regarding the intervention study, it is expected that there will be an improvement in eating behavior; weight, weight regain reversal, self-image classification; in the quality of life; and in the levels of mindfulness, self-pity and anxiety of these patients. This study hopes to gather preliminary evidence on the effectiveness of mindfulness and compassion training for the adjuvant treatment of weight regain in post-bariatric patients.

DETAILED DESCRIPTION:
This is a randomized intervention study with four protocols (MBHP + TAU, ABCT + TAU and TAU) to be performed with patients who underwent at least two years of bariatric surgery in 2012 and 2017 in a private clinic for obesity treatment in Uberlândia - Minas Gerais and who had regained weight. The study site will consist of a private obesity treatment clinic located in Uberlândia - Minas Gerais, founded in 2011 and which has performed approximately 5000 gastroplasty. It has an integrated multidisciplinary team composed of 4 doctors (2 bariatric surgeons, 1 gastroenterologist and 1 pulmonologist), 3 nutritionists, 2 psychologists and 1 nurse, who values both the patient's physical and mental health. Participants will be the adult patients who underwent gastroplasty (sleeve gastrectomy or Roux-en-Y gastric Bypass) from the clinic. All patients will be invited to participate in two support group meetings - usual treatment (TAU) - provided by the bariatric surgery clinic of this study. Subsequently, participants will be allocated into four groups, MBHP, ABCT and TAU. Participants of the MBHP and ABCT groups will also be invited to participate in the respective intervention protocols. Participants who remain in the TAU group after phase 2 will be invited to participate in the intervention group that has the most benefit to patients. All travel / travel expenses incurred by participants will be reimbursed. Measurements and evaluations will be performed 1 week before baseline (T0), after 2 months, post-intervention period (T1) and 6 months after intervention (T2). The following interventions will be performed live and online as follows: Patients will meet at the Bariatric Surgery Clinic of that study and instructors will be available for each session on scheduled days and times. The MBHP model is a program designed to address universal human vulnerabilities, not focusing on any specific health condition. Structured and developed over eight weeks (8 sessions), participants meet weekly for an average of 2 hours to experience the techniques and conceptual learning about mindfulness, and can be adapted to one or 1.5 hour sessions. to be applicable within the contexts of health, education and organizations. Participants are also given suggested activities to be implemented in a home or work setting on a daily basis, lasting an average of 15-20 minutes and up to 45 minutes for more motivated and adherent participants. They are instructed to seek to incorporate the idea of mindfulness into their daily lives (activity called informal practice), making routine activities somehow an opportunity to use the state of mindfulness. The main mindfulness techniques used are mindfulness breathing practice, body scanning (technique relatively similar to progressive muscle relaxation), mindfulness walking, mindfulness movements, in which lightweight body activities are used. be performed by individuals with different levels of ability and with physical limitations. One of the sessions (sixth session) is held in silence, with the purpose of deepening the practices 37 The ABCT is a program based on one of the fundamental psychological constructs that explain the interpersonal relationships of individuals, attachment styles. It lasts 8 weeks in which participants meet for 2 or 2.5 hours in each meeting. ABCT teaches formal (sitting meditation) and informal (during daily life) self-compassion. There are experimental exercises and discussion periods in each session, as well as homework, to help participants learn how to be kind to themselves. The control group (TAU) and the other participants will receive the usual treatment for post-bariatric patients of the clinic in question, which is the participation in support groups offered by the bariatric surgery clinic with capacity for 40 participants, monthly frequency and duration of 2 hours In these meetings there is always the presence of a surgeon, a psychologist and another guest professional (endocrinologist, nutritionist, speech therapist or dentist), who give a thematic lecture and then there is the opening space for doubts and exchange of experiences. All protocol instructors will be certified by internationally validated mindfulness institutions with extensive experience in conducting MBHP and ABCT groups. The methodological procedures of the present work were prepared within the fundamental ethical and scientific procedures, as provided for in Resolution No. 466 of December 12, 2012 of the National Health Council of Ministry of Health, being approved by the Research Ethics Committee (CEP), by protocol 18529519.5.0000.5505. The primary outcome will be the modification of eating behavior (Three factor eating questionnaire and Repetitive Eating Questionnaire). Secondary outcomes will be the improvement in quality of life (Bariatric analysis and reporting outcome system), body image (Brazilian Silhouette Scales for adults and children) and better weight management (weight maintenance or reduction). And the explanatory variables are: Level of Mindful Attention Awareness Scale, Self-compassion Scale, anxiety, greater adherence to sessions and higher frequency of formal practice throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Weight regain ≥ 5% of the minimum achieved postoperatively
* Literate
* Consent to Randomization

Exclusion Criteria:

* Use of weight loss medication;
* Pregnancy;
* Substance abuse (alcohol or drugs);
* State of acute depression (<6 months of diagnosis), diagnosed schizophrenia or psychotic disorders, use of drugs that cause cognitive loss of attention and concentration (such as potent anxiolytic medications)
* Prior mindfulness, meditation, yoga or similar practices in the last 6 months (with formal practice at least once a week).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 456 (Estimated)
Dates: Start 2019-11-05 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Mean Change from Baseline in food behavior scores | T0 (baseline), T1(end of treatment at 8 weeks) and T2 (six months after the end of treatment)
  The Three factor eating questionnaire (1-100: higher scores indicate more uncontrolled, restraint and emotional eating. Scores closest to 100 indicate a worse outcome) and Repetitive eating questionnaire (higher scores indicate more repetitive eating. Scores closest to 6 indicate a worse outcome)

SECONDARY OUTCOMES:
Mean Change from Baseline in quality of life level | T0 (baseline), T1(end of treatment at 8 weeks) and T2 (six months after the end of treatment)
  Bariatric analysis and reporting outcome system
Change from Baseline in self perception body image | T0 (baseline), T1(end of treatment at 8 weeks) and T2 (six months after the end of treatment)
  Brazilian Silhouette Scales for Adults (1-15: higher scores indicate higher perceived Body Mass Index, which is neither good nor bad).
Weight change | T0 (baseline), T1(end of treatment at 8 weeks) and T2 (six months after the end of treatment)
  measure of weight

OTHER OUTCOMES:
Change from Baseline in Mindfulness score | T0 (baseline), T1(end of treatment at 8 weeks) and T2 (six months after the end of treatment)
  Mindful Attention Awareness Scale
Change from Baseline in Self-compassion score | T0 (baseline), T1(end of treatment at 8 weeks) and T2 (six months after the end of treatment)
  Self-compassion Scale (12-60: higher scores indicate more self-compassion. Scores closest to 60 indicate a better outcome)
Change from Baseline in anxiety score | T0 (baseline), T1(end of treatment at 8 weeks) and T2 (six months after the end of treatment)
  Mindful Attention Awareness Scale (1-6: higher scores indicate more mindfuness. Scores closest to 6 indicate a better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Erika BS Porto, Master, Principal Investigator — Federal Univesity of São Paulo
Locations (1):
- Centro Mente Aberta de Mindfulness e Promoção de Saúde, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared by research gate
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: December, 2021. Will be available for 2 years
Access Criteria: Access will be granted to those researchers who are interested in developing studies with objectives similar to this research.

REFERENCES:
- [Background] WHO. Fiscal policies for diet and the prevention of noncommunicable diseases. WHO Reg Off Eur. 2015;(May):36. http://www.who.int/dietphysicalactivity/publications/fiscal-policies-diet-prevention/en/.
- [Background] Instituto Brasileiro de Geografia e Estatística. Antropometria e estado nutricional de crianças, adolescentes e adultos no Brasil. 2009;1:45.
- [Background] BRASIL. Vigitel Brasil 2017: Vigilância de Fatores de Risco e Proteção Para Doenças Crônicas Por Inquérito Telefônico : Estimativas Sobre Frequência e Distribuição Sociodemográfica de Fatores de Risco e Proteção Para Doenças Crônicas Nas Capitais Dos 26 Estados B. Brasília: Ministério da Saúde; 2018. http://bvsms.saude.gov.br/bvs/publicacoes/vigitel_brasil_2017_vigilancia_fatores_. Accessed September 12, 2018.
- [Background] Adams TD, Gress RE, Smith SC, Halverson RC, Simper SC, Rosamond WD, Lamonte MJ, Stroup AM, Hunt SC. Long-term mortality after gastric bypass surgery. N Engl J Med. 2007 Aug 23;357(8):753-61. doi: 10.1056/NEJMoa066603. PMID 17715409
- [Background] Karmali S, Brar B, Shi X, Sharma AM, de Gara C, Birch DW. Weight recidivism post-bariatric surgery: a systematic review. Obes Surg. 2013 Nov;23(11):1922-33. doi: 10.1007/s11695-013-1070-4. PMID 23996349
- [Background] Mechanick JI, Youdim A, Jones DB, Garvey WT, Hurley DL, McMahon MM, Heinberg LJ, Kushner R, Adams TD, Shikora S, Dixon JB, Brethauer S; American Association of Clinical Endocrinologists; Obesity Society; American Society for Metabolic & Bariatric Surgery. Clinical practice guidelines for the perioperative nutritional, metabolic, and nonsurgical support of the bariatric surgery patient--2013 update: cosponsored by American Association of Clinical Endocrinologists, the Obesity Society, and American Society for Metabolic & Bariatric Surgery. Endocr Pract. 2013 Mar-Apr;19(2):337-72. doi: 10.4158/EP12437.GL. PMID 23529351
- [Background] Pope GD, Finlayson SR, Kemp JA, Birkmeyer JD. Life expectancy benefits of gastric bypass surgery. Surg Innov. 2006 Dec;13(4):265-73. doi: 10.1177/1553350606296324. PMID 17227925
- [Background] Sjostrom L, Lindroos AK, Peltonen M, Torgerson J, Bouchard C, Carlsson B, Dahlgren S, Larsson B, Narbro K, Sjostrom CD, Sullivan M, Wedel H; Swedish Obese Subjects Study Scientific Group. Lifestyle, diabetes, and cardiovascular risk factors 10 years after bariatric surgery. N Engl J Med. 2004 Dec 23;351(26):2683-93. doi: 10.1056/NEJMoa035622. PMID 15616203
- [Background] Angrisani L, Santonicola A, Iovino P, Formisano G, Buchwald H, Scopinaro N. Bariatric Surgery Worldwide 2013. Obes Surg. 2015 Oct;25(10):1822-32. doi: 10.1007/s11695-015-1657-z. PMID 25835983
- [Background] Magro DO, Ueno M, Coelho-Neto JS, Callejas-Neto F, Pareja JC, Cazzo E. Long-term weight loss outcomes after banded Roux-en-Y gastric bypass: a prospective 10-year follow-up study. Surg Obes Relat Dis. 2018 Jul;14(7):910-917. doi: 10.1016/j.soard.2018.03.023. Epub 2018 Mar 26. PMID 29706496
- [Background] Fried M, Yumuk V, Oppert JM, Scopinaro N, Torres A, Weiner R, Yashkov Y, Fruhbeck G; International Federation for Surgery of Obesity and Metabolic Disorders-European Chapter (IFSO-EC); European Association for the Study of Obesity (EASO); European Association for the Study of Obesity Obesity Management Task Force (EASO OMTF). Interdisciplinary European guidelines on metabolic and bariatric surgery. Obes Surg. 2014 Jan;24(1):42-55. doi: 10.1007/s11695-013-1079-8. PMID 24081459
- [Background] Nedelcu M, Khwaja HA, Rogula TG. Weight regain after bariatric surgery-how should it be defined? Surg Obes Relat Dis. 2016 Jun;12(5):1129-1130. doi: 10.1016/j.soard.2016.04.028. Epub 2016 Apr 29. No abstract available. PMID 27350180
- [Background] Velapati SR, Shah M, Kuchkuntla AR, Abu-Dayyeh B, Grothe K, Hurt RT, Mundi MS. Weight Regain After Bariatric Surgery: Prevalence, Etiology, and Treatment. Curr Nutr Rep. 2018 Dec;7(4):329-334. doi: 10.1007/s13668-018-0243-0. PMID 30168043
- [Background] Palmeira L, Cunha M, Pinto-Gouveia J. Processes of change in quality of life, weight self-stigma, body mass index and emotional eating after an acceptance-, mindfulness- and compassion-based group intervention (Kg-Free) for women with overweight and obesity. J Health Psychol. 2019 Jul;24(8):1056-1069. doi: 10.1177/1359105316686668. Epub 2017 Jan 10. PMID 28810375
- [Background] Paul L, van der Heiden C, Hoek HW. Cognitive behavioral therapy and predictors of weight loss in bariatric surgery patients. Curr Opin Psychiatry. 2017 Nov;30(6):474-479. doi: 10.1097/YCO.0000000000000359. PMID 28795980
- [Background] Lynch AI, McGowan E, Zalesin KC. "Take Me through the History of Your Weight": Using Qualitative Interviews to Create Personalized Weight Trajectories to Understand the Development of Obesity in Patients Preparing for Bariatric Surgery. J Acad Nutr Diet. 2018 Sep;118(9):1644-1654. doi: 10.1016/j.jand.2017.12.008. Epub 2018 Mar 16. PMID 29551398
- [Background] Heriseanu AI, Hay P, Corbit L, Touyz S. Grazing in adults with obesity and eating disorders: A systematic review of associated clinical features and meta-analysis of prevalence. Clin Psychol Rev. 2017 Dec;58:16-32. doi: 10.1016/j.cpr.2017.09.004. Epub 2017 Sep 15. PMID 28988855
- [Background] Kahl KG, Winter L, Schweiger U. The third wave of cognitive behavioural therapies: what is new and what is effective? Curr Opin Psychiatry. 2012 Nov;25(6):522-8. doi: 10.1097/YCO.0b013e328358e531. PMID 22992547
- [Background] Mason AE, Epel ES, Kristeller J, Moran PJ, Dallman M, Lustig RH, Acree M, Bacchetti P, Laraia BA, Hecht FM, Daubenmier J. Effects of a mindfulness-based intervention on mindful eating, sweets consumption, and fasting glucose levels in obese adults: data from the SHINE randomized controlled trial. J Behav Med. 2016 Apr;39(2):201-13. doi: 10.1007/s10865-015-9692-8. Epub 2015 Nov 12. PMID 26563148
- [Background] Christensen BJ, Iepsen EW, Lundgren J, Holm L, Madsbad S, Holst JJ, Torekov SS. Instrumentalization of Eating Improves Weight Loss Maintenance in Obesity. Obes Facts. 2017;10(6):633-647. doi: 10.1159/000481138. Epub 2017 Dec 6. PMID 29207396
- [Background] Mitchell JE, Christian NJ, Flum DR, Pomp A, Pories WJ, Wolfe BM, Courcoulas AP, Belle SH. Postoperative Behavioral Variables and Weight Change 3 Years After Bariatric Surgery. JAMA Surg. 2016 Aug 1;151(8):752-7. doi: 10.1001/jamasurg.2016.0395. PMID 27096225
- [Background] Warren JM, Smith N, Ashwell M. A structured literature review on the role of mindfulness, mindful eating and intuitive eating in changing eating behaviours: effectiveness and associated potential mechanisms. Nutr Res Rev. 2017 Dec;30(2):272-283. doi: 10.1017/S0954422417000154. Epub 2017 Jul 18. PMID 28718396
- [Background] Neff K. Self-Compassion: An Alternative Conceptualization of a HealthyAttitudeToward Oneself. Self Identity. 2003;2:85-101. doi:10.1080/15298860390129863
- [Background] Adams CE, Leary MR. ADAMS AND LEARY SELF-COMPASSIONATE EATING ATTITUDES PROMOTING SELF-COMPASSIONATE ATTITUDES TOWARD EATING AMONG RESTRICTIVE AND GUILTY EATERS. J Soc Clin Psychol. 2007;26(10):1120-1144. https://www.weightcrafters.com/adams-leary-eating-attitudes.pdf. Accessed June 3, 2018.
- [Background] Neff KD, Germer CK. A pilot study and randomized controlled trial of the mindful self-compassion program. J Clin Psychol. 2013 Jan;69(1):28-44. doi: 10.1002/jclp.21923. Epub 2012 Oct 15. PMID 23070875
- [Background] Mason AE, Epel ES, Aschbacher K, Lustig RH, Acree M, Kristeller J, Cohn M, Dallman M, Moran PJ, Bacchetti P, Laraia B, Hecht FM, Daubenmier J. Reduced reward-driven eating accounts for the impact of a mindfulness-based diet and exercise intervention on weight loss: Data from the SHINE randomized controlled trial. Appetite. 2016 May 1;100:86-93. doi: 10.1016/j.appet.2016.02.009. Epub 2016 Feb 8. PMID 26867697
- [Background] Palmeira L, Pinto-Gouveia J, Cunha M. Exploring the efficacy of an acceptance, mindfulness & compassionate-based group intervention for women struggling with their weight (Kg-Free): A randomized controlled trial. Appetite. 2017 May 1;112:107-116. doi: 10.1016/j.appet.2017.01.027. Epub 2017 Jan 21. PMID 28119138
- [Background] Spadaro KC, Davis KK, Sereika SM, Gibbs BB, Jakicic JM, Cohen SM. Effect of mindfulness meditation on short-term weight loss and eating behaviors in overweight and obese adults: A randomized controlled trial. J Complement Integr Med. 2017 Dec 5;15(2):/j/jcim.2018.15.issue-2/jcim-2016-0048/jcim-2016-0048.xml. doi: 10.1515/jcim-2016-0048. PMID 29211681
- [Background] Chacko SA, Yeh GY, Davis RB, Wee CC. A mindfulness-based intervention to control weight after bariatric surgery: Preliminary results from a randomized controlled pilot trial. Complement Ther Med. 2016 Oct;28:13-21. doi: 10.1016/j.ctim.2016.07.001. Epub 2016 Jul 12. PMID 27670865
- [Background] Maia RP, Silva PCC da, Duarte ACS, Costa RM da. Avaliação Do Perfil Nutricional E Qualidade De Vida Após Realização De Cirurgia Bariátrica Em Um Hospital Público De Goiânia, Brasil. DEMETRA Aliment Nutr Saúde. 2018;13(1):147-164. doi:10.12957/demetra.2018.27515
- [Background] Natacci LC, Júnior MF. The three factor eating questionnaire - R21: Tradução para o português e aplicação em mulheres brasileiras. Rev Nutr. 2011;24(3):383-394. doi:10.1590/S1415-52732011000300002
- [Background] Conceicao EM, Mitchell JE, Machado PPP, Vaz AR, Pinto-Bastos A, Ramalho S, Brandao I, Simoes JB, de Lourdes M, Freitas AC. Repetitive eating questionnaire [Rep(eat)-Q]: Enlightening the concept of grazing and psychometric properties in a Portuguese sample. Appetite. 2017 Oct 1;117:351-358. doi: 10.1016/j.appet.2017.07.012. Epub 2017 Jul 13. PMID 28712976
- [Background] Oria HE, Moorehead MK. Bariatric analysis and reporting outcome system (BAROS). Obes Surg. 1998 Oct;8(5):487-99. doi: 10.1381/096089298765554043. PMID 9819079
- [Background] Kakeshita IS, Silva AIP, Zanatta DP, Almeida SS. Construção e fidedignidade teste-reteste de escalas de silhuetas brasileiras para adultos e crianças. Psicol Teor e Pesqui. 2010;25(2):263-270. doi:10.1590/s0102-37722009000200015
- [Background] Marcolino JA, Mathias LA, Piccinini Filho L, Guaratini AA, Suzuki FM, Alli LA. Hospital Anxiety and Depression Scale: a study on the validation of the criteria and reliability on preoperative patients. Rev Bras Anestesiol. 2007 Feb;57(1):52-62. doi: 10.1590/s0034-70942007000100006. English, Portuguese. PMID 19468618
- [Background] nstituto Brasileiro de Geografia e Estatística. Sinopse Do Censo Demográfico 2010. Rio de Janeiro; 2011. www.ibge.gov.br/cidade@.
- [Background] Campayo MD e javier G. Manual Prático Mindfulness Curiosidade e Aceitação. 3a. São Paulo; 2015.
- [Background] Garcia-Campayo J, Demarzo M. Attachment-based compassion therapy Telessaúde em APS View project (C)BT vs. Relaxation in Anxiety Disorders: a meta-analysis View project. mindfulness et compassion. 2016;1:68-74. doi:10.1016/j.mincom.2016.10.004
- [Background] Luiza Akiko Komura Hoga Ana Luiza Vilela Borges C, Edição São Paulo a. Pesquisa Empírica Em Saúde: Guia Prático Par Iniciantes.; 2016. http://www.ee.usp.br/cartilhas/pesquisa_empirica_saude_2016.pdf. Accessed July 23, 2018.
- [Derived] Porto EBS, Montero-Marin J, Quadros LG, Kristeller J, Sarubbi Junior V, Mattar LA, Garcia-Campayo J, Demarzo M. Mindfulness and compassion-based programs on eating behavior of post-bariatric surgery patients: A two phased clinical trial protocol. MethodsX. 2024 Aug 9;13:102885. doi: 10.1016/j.mex.2024.102885. eCollection 2024 Dec. PMID 39253004